CLINICAL TRIAL: NCT06688695
Title: Intervention for Neurodevelopmental Support in Preterm Infants Using Responsive Parenting and E-health (INSPIRE)
Brief Title: Intervention for Neurodevelopmental Support in Preterm Infants Using Responsive Parenting and E-health
Acronym: INSPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EPM Dnr 2024-03048-01
Record Dates: First submitted 2024-10-03; First posted 2024-11-14 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Premature Infant; Premature Babies
Keywords: Early intervention; Responsive parenting; E-health; Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controll group (No Intervention): Standard care
- INSPIRE-intervention (Other): Intervention group, recieving the INSPIRE-intervention
  Interventions: Behavioral: Neurodevelopmental support

INTERVENTIONS:
Behavioral: Neurodevelopmental support — The Intervention for Neurodevelopmental Support in Preterm Infants using Responsive parenting and E-health (INSPIRE) aims to support the infant's neurodevelopment by supporting the parents to develop a responsive approach. The intervention will enhance the infant's social and environmental interactions, focusing on developing both the infant's and parent's strengths, seeking opportunities instead of problems in behaviour, enhancing mutually satisfying interaction and parental empowerment.
  Arms: INSPIRE-intervention

SUMMARY:
Research problem and specific questions More than 1000 very preterm infants (< 32 weeks) are born every year in Sweden. They are at high risk of neurodevelopmental disabilities and mental illness throughout the lifespan.

The overall purpose is to develop and evaluate a novel e-health intervention aimed at improving neurodevelopment (cognitive, motor, feeding, language, socio-emotional) of very preterm infants by supporting responsive parenting behaviours.

The primary research question is whether the intervention improves child neurodevelopment up to 2 years.

Further research questions relate to the emotional availability of parents and children, parental stress and overall experience as well as effects on health inequalities and gender effects.

Data and method Using a multi-professional approach, the study team have developed a post-discharge "Intervention for Neurodevelopmental Support in Preterm Infants using Responsive parenting and E-health" (INSPIRE). Parents of very preterm infants will be included in the program at hospital discharge and will receive the intervention in 18 sessions over a two year period.

The study team have assessed feasibility and refined the intervention in a pilot study including 9 families. This autumn, a randomized clinical trial will be performed to evaluate efficiency: Families will be randomized to the INSPIRE program or standard care. Follow-up and assessment of children (and parents) across a range of crucial domains will be performed up to at least 2 years of age.

Societal relevance and utilisation The project will be the first in the world to use a digital e-health solution with video interaction to deliver a post discharge parental support intervention to parents of very preterm infants. The project has great potential to reduce the risk of cognitive impairment, behavioral problems, mental illness and eating disorders in these high risk children, as well as improving mental health and well-being in the parents. Parents of preterm infants are involved as co-creators in developing and evaluating the program.

Plan for project realization Currently, there is no similar post-discharge program available. Based on the results, the study team aim to implement a sustainable, nationwide, post-discharge e-health intervention program to improve health in very preterm-born children and their parents, which will also reduce health inequality by ensuring the availability of high-quality support to families living far away from highly specialized health care facilities

ELIGIBILITY:
Inclusion Criteria:

* Infant born before 32 GV, or with birth weight under 1500 gr.

Exclusion Criteria:

* Parent(s) younger than 18 ya.
* Chromosomal abnormalities, congenital syndromes that may affect the child's development.
* Parents unable to understand Swedish.
* Parents with severe mental illness or a physical medical condition requiring extensive inpatient care.
* Families without a stable living situation, such as parental substance abuse, homelessness, or family living under threat of deportation from Sweden.
* Families that have previously participated in the INSPIRE study or the INSPIRE pilot study.

Ages: 0 Months to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Bayley Scales of Infant Development (BSID IV) | 24 months corrected age
  Bayley Scales of Infant Development (BSID IV) is a test administered by a psychologist for assessment of general neurodevelopment (cognitive, language and motor) at 24 months corrected age (primary outcome)

SECONDARY OUTCOMES:
Alberta infant motor scale (AIMS) | 6 months corrected age.
  Alberta infant motor scale is a test performed by a physiotherapist, based on live observation or a video recording of the infant. We will use video recordings.
Peabody Developmental Motor Scales (PDMS-2) | 24 months corrected age.
  Peabody Developmental Motor Scales (PDMS-2) is a test, administered by a physiotherapist, to assess motor function.
Wechsler Preschool and Primary Scale of Intelligence, 4th Edition (WPPSI IV) | 5,5 years of age
  Wechsler Preschool and Primary Scale of Intelligence, 4th Edition (WPPSI IV) is a test performed by a psychologist for assessment of cognitive development at 5.5 years of age.
Movement ABC | 5,5 years of age
  Movement ABC is a test administered by a physiotherapist for assessment of motor development at 5.5 years of age.
Strengths and Difficulties Questionnaire (SDQ) | 24 months corrected age, 36 months of age and 5,5 years of age
  Strengths and Difficulties Questionnaire (SDQ) is a parental questionnaire for assessment of behavioural problems
The Infant Toddler Checklist (ITC) | 18 months corrected age
  The Infant Toddler Checklist (ITC) is a questionnaire/method to assess early language development
The MacArthur-Bates Communicative Development Inventories (MB-CDIs) | 12 and 18 months corrected age.
  The MacArthur-Bates Communicative Development Inventories (MB-CDIs) is a questionnaire/method to assess early language development.
"Jollerobservation" | 12 months corrected age.
  "Jollerobservation" is a Swedish standardised protocol for observation of babbling. The observation is performed by a speech- and language pathologist.
The Montreal Children's Hospital Feeding Scale | 12 months corrected age.
  The Montreal Children's Hospital Feeding Scale are a questionnaire that will be used for assessment of feeding development.
The Emotional Availability Scale (EAS) | 12 months corrected age and 24 months corrected age.
  The Emotional Availability Scale (EAS) is an observational coding system to assess emotional availability during caregiver-infant interactions regarding both the parent and the child
The Parental Reflective Functioning Questionnaire (PRFQ) | At enrollment (at 38-42 weeks postmenstrual age), at 12 months corrected age, 24 months corrected age, and 36 months of age and 5,5 years of age.
  The Parental Reflective Functioning Questionnaire (PRFQ) will be used to assess parents reflective functioning regarding their child's emotional needs
Modified Checklist for Autism in Toddlers (M-CHAT | 24 months corrected age
  Modified Checklist for Autism in Toddlers (M-CHAT) is a parental questionnaire for assessment of early signs of autism
The Reynell Developmental Language Scales IV (RDLS IV) | 36 months of age.
  The Reynell Developmental Language Scales IV (RDLS IV) will be used for detailed assessment of language development.
Ages and Stages Questionnaire (ASQ) | 24 months corrected age
  Ages and Stages Questionnaire (ASQ) is a parental questionnaire for assessment of general neurodevelopment
Swedish Parenthood Stress Questionnarie (SPSQ) | At enrollment (at 38-42 weeks postmenstrual age), at 12 months corrected age, 24 months corrected age, and 36 months of age and 5,5 years of age.
  Swedish Parenthood Stress Questionnarie (SPSQ) is a questionnaire that measures stress.
Resilience Scale (RES) | At enrollment (at 38-42 weeks postmenstrual age), at 12 months corrected age, 24 months corrected age, and 36 months of age and 5,5 years of age.
  Resilience Scale (RES) is a questionnaire that measures resilience.
Parental Self-Efficacy Scale (PSE) | At enrollment (at 38-42 weeks postmenstrual age), at 12 months corrected age, 24 months corrected age, and 36 months of age and 5,5 years of age.
  Parental Self-Efficacy Scale (PSE) is a questionnaire that measures parental self efficacy.
The Hospital Anxiety and Depression scale (HAD) | At enrollment (at 38-42 weeks postmenstrual age), at 12 months corrected age and 5,5 years of age.
  The Hospital Anxiety and Depression scale (HAD) is a questionnaire that measures anxiety and depression. It will be used to assess parental mental health.
The State-Trait Anxiety Inventory (STAI) | At enrollment (at 38-42 weeks postmenstrual age), at 12 months corrected age and 5,5 years of age.
  The State-Trait Anxiety Inventory (STAI) is a questionnaire that measures anxiety. It will be used to assess parental mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Domellöf, Professor, Study Director — Umeå universitet
Locations (7):
- Sweden (7):
  - Falu County Hospital, Falun, Dalarna County
  - Östersund Hospital, Östersund, Jämtland Härjedalen
  - Sunderby Hospital, Södra Sunderbyn, Norrbotten County
  - Karlstad Hospital, Karlstad, Värmland County
  - Umeå university hospital, Umeå, Västerbotten County
  - Sundsvall Hospital, Sundsvall, Västernorrland County
  - Örebro University Hospital, Örebro, Örebro County

IPD SHARING:
Plan to Share IPD: No